CLINICAL TRIAL: NCT06280378
Title: A Phase I/II Clinical Study Evaluating the Safety and Efficacy of KL003 Cell Injection in Transfusion-dependent Β-thalassemia
Brief Title: Β-Thalassemia Treatment with KL003 Cell Injection
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kanglin Biotechnology (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-KL003-003/01
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-04

CONDITIONS: Transfusion-dependent Beta-Thalassemia
Keywords: gene therapy; lentiviral vector; KL003 cell injection; transfusion-dependent β-thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KL003 Cell Injection Drug Product (Experimental): Transplant of auto-HSC transduced with lentiviral vector encoding βA-T87Q-globin gene
  Interventions: Drug: KL003 Cell Injection Drug Product

INTERVENTIONS:
Drug: KL003 Cell Injection Drug Product — Administered by intravenous infusion after myeloablative conditioning with busulfan.

SUMMARY:
This is a non-randomized, open label, single-dose study in up to 41 participants with β-thalassemia major. The goal of this clinical trial is to evaluate the safety and efficacy of KL003 cell injection in subjects with β-thalassemia major.

DETAILED DESCRIPTION:
This is a single-arm, multi-site, single-dose, Phase 1/2 study to assess KL003 Cell Injection in up to 41 participants with transfusion-dependent β-thalassemia (TDT) who are ≥3 and ≤35 years of age. KL003 Cell Injection is autologous CD34+ stem cells transduced Ex Vivo with a lentiviral Vector encoding βA-T87Q-Globin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age between 3-35 years;
* Diagnosis of transfusion-dependent β-thalassemia and a history of at least 100 mL/kg/year of pRBCs or ≥8 transfusions of pRBCs per year for the prior 2 years;
* Karnofsky performance status ≥70 for participants≥16 years of age; Lansky performance status of ≥70 for participants<16 years of age;
* Eligible to undergo auto-HSCT;
* Willing and able to follow the research procedures and conditions, with good compliance;
* Willing to receive at least the 2 years follow-up;
* Participant and/or legal guardians voluntarily participated in this clinical trial and signed the informed consent form.

Exclusion Criteria:

* Diagnosis of composite α thalassemia;
* Prior receipt of gene therapy or allo-HSCT;
* Meet the criteria for allo-HSCT and with an identified willing donor with full HLA match;
* Participants with severe iron overload at the time of screening;
* Presence of unusual antibody of red blood cell antigens or tested positive for platelet antibody;
* Known allergy to clinical trial drug (plerixafor or G-CSF or busulfan) or ingredient(DMSO etc.);
* Clinically significant and active bacterial, viral, fungal, or parasitic infection as determined by the clinical investigator;
* Subjects positive with the following etiological tests: human immunodeficiency virus(HIV-1-2),human cytomegalovirus (HCMV-DNA),EB virus（EBV-DNA）,HBV (HBsAg/HBV-DNA positive),HCV antibody (HCV-Ab), Human T-lymphotropic virus antibody (HTLV-Ab), Treponema pallidum antibody (TP-Ab);
* Uncorrectable coagulation dysfunction or history of severe bleeding disorder;
* History of major organ damage including:

  1. Liver function test suggest AST or ALT levels >3× upper limit of normal（ULN）;
  2. Total serum bilirubin value>2.5×ULN;if combined with Gilbert syndrome, total bilirubin>3×ULN and direct bilirubin value>2.5×ULN;
  3. Left ventricular ejection fraction <45%;
  4. Baseline calculated eGFR<60mL/min/1.73m2;
  5. Pulmonary function:FEV1/FVC<60% and/or diffusion capacity of carbon monoxide (DLco) <60% of prediction;

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
KL003 engraftment | From time of KL003 infusion through Month 2
  Proportion of participants with successful engraftment within 42 days after KL003 infusion.
Engraftment time of neutrophil and platelet | From time of KL003 infusion through Month 24
  Neutrophil engraftment was defined as the first day when neutrophils ≥ 0.5×10^9/L for 3 consecutive days; Platelet engraftment was defined as the first the first day of platelet count ≥ 20.0×10^9/L for 7 consecutive days with no platelet transfusions.
Overall Survival | From time of KL003 infusion through Month 24
  Overall survival was defined as time from date of KL003 infusion to date of death.
The number, frequency and severity of adverse events (AE) within 1 year after infusion of KL003 drug products | From time of KL003 infusion through Month 24
  Frequency and severity of AEs & SAEs identified according to NCI CTCAE 5.0
Clonal dominance or secondary tumors caused by lentiviral vector insertional-mutation | From time of KL003 infusion through Month 24
  Clonal dominance was defined as an ISA result greater than 90% of the total insertion sites (IS) at any time
Numbers of Participants With Vector-Derived Replication-Competent Lentivirus (RCL) | From time of KL003 infusion through Month 24
  Peripheral blood samples were analyzed for detection of RCL

SECONDARY OUTCOMES:
The proportion of participants achieved Transfusion Independence (TI)for at least 6 months | From time of KL003 infusion through Month 24
  TI 6 is defined as Hb ≥ 90.0 g/L after reinfusion and without disease-related routine blood transfusion for 6 months
The proportion of participants achieved TI 12 | From time of KL003 infusion through Month 24
  TI 12 is defined as Hb ≥ 90.0 g/L after reinfusion and without disease-related routine blood transfusion for 12 months
The start time of Transfusion Independence (TI) after KL003 infusion | From time of KL003 infusion through Month 24
  The TI start time is defined as the first day of treated participants with transfusion-dependent β-thalassemia (TDT) who achieved transfusion independence.
Total Hb and the vector-derived HbA^T87Q | From time of KL003 infusion through Month 24
  The total Hb is measured by routine blood test, Therapeutic globin expression was measured by HbA^T87Q in peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Haoquan Wu, PhD, Study Director — R&D Kanglin Biotech
Locations (2):
- China (2):
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No